CLINICAL TRIAL: NCT03520335
Title: Implementation of Finnish Prehospital Stroke Scale (FPSS) to Emergency Medical Services - a Prospective, Multi-centre Study
Brief Title: Implementation of Finnish Prehospital Stroke Scale to Emergency Medical Services
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Central Finland Hospital District (Other); Vaasa Central Hospital, Vaasa, Finland (Other); Seinajoki Central Hospital (Other); Satakunta Central Hospital (Other); PaijatHame Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R18010
Record Dates: First submitted 2018-04-25; First posted 2018-05-09 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Recognition of Thrombectomy Candidate
Keywords: stroke; conjugated eye deviation; prehospital; stroke scale; large vessel occlusion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators have developed a simple prehospital stroke scale (FPSS), containing 5 dichotomized items to recognize both large and small artery thrombi of the brain. FPSS is implemented to both emergency medical services and later, to emergency response centers. The efficacy of the scale and possible improvement of both the patient flow and treatment results will be evaluated.

DETAILED DESCRIPTION:
Finnish Prehospital Stroke Scale, FPSS, was developed for prehospital setting for prediction of large vessel occlusions (LVOs) and stroke in common. It contains four stroke signs used universally in emergency medical services (EMSs) and emergency response centers (ERCs): 1) facial weakness, 2) extremity weakness, 3) speech disturbance, 4) visual disturbance. Additionally, it contains only one item 5) conjugated gaze deviation, while all the items are presented in dichotomized form. In an earlier, retrospective cohort of 856 code stroke patients, the sensitivity of FPSS for LVOs was highest for thrombi of areas with the documented cost effectiveness of endovascular treatment: internal carotid artery (ICA) and M1 segment of middle cerebral artery (72 % and 82 %). The overall specificity of FPSS for the LVOs was 91 %. For its simplicity it is easy to implement in EMS and ERC as a single score predicting both thrombolysis and thrombectomy candidates.

In the present study accuracy of FPSS will be studied prospectively. FPSS is launched 5/18 in EMS in an area with a population of more than a million, containing districts of five central hospitals capable for thrombolysis and one university hospital capable for endovascular treatment. During 2019-20 FPSS will be launched in two ERCs triaging stroke patients in the study area.

The hypotheses that are tested are:

1. FPSS is accurate to detect ICA and M1 thrombi in EMS setting
2. The use of FPSS shortens door-in-door-out (DIDO) delay patients arriving to central hospitals and redirected to university hospital for thrombectomy.
3. The use of FPSS aids to triage LVO-patients straight to a center capable for thrombectomy
4. FPSS is accurate in the detection of ICA and M1 thrombi in ERC setting
5. The effect of fluent triage of LVO is seen in overall shortened recanalization delay and better outcomes as lower modified Rankin Scores (mRS) in 3 months control compared recanalization delays and 3 month mRS during the pre-implementation period.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischaemic stroke
* Prehospital susipicion of large vessel occlusion

Exclusion Criteria:

- Stroke mimic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with acute stroke in a population of 1 million
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 3 years
  Accuracy of Finnish Prehospital Stroke Scale used in prehospital settingto detect a large vessel occlusion
  Finnish Prehospital Stroke Scale (FPSS) includes the following items:
  Facial droop 0-1, Weakness of one or more extremities 0-1, Difficulty of understand or produce speech, including slurring 0-1, Field cut of visus or blindness 0-1, Partial or fixed gaze or head deviation away from the paretic side 0 or 4. Total points 1-4 predicts non-LVO, ≥ 5 predicts LVO 0-8 (non-LVO= small or medium-sized vessel occlusion; iv-thrombolysis candidate; LVO= large vessel occlusion; endovascular treatment candidate)

SECONDARY OUTCOMES:
90 day survival | 3 years
  90 day survival
90 day modified Rankin score | 3 years
  90 day modified Rankin score
Onset to treatment time | 3 years
  Onset to treatment time

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided